CLINICAL TRIAL: NCT04207281
Title: Honey to Improve Sleep Quality: a Randomized, Double-blind Trial
Brief Title: Honey to Improve Sleep Quality
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Jane Alcorn, Dean and Professor of Pharmacy and Nutrition, University of Saskatchewan
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Bio-1666
Record Dates: First submitted 2019-12-18; First posted 2019-12-20 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Poor Quality Sleep

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Honey (Active Comparator): Raw honey (1.5 tablespoons)
  Interventions: Dietary Supplement: Raw Honey; Dietary Supplement: Comparator
- Comparator (Placebo Comparator): Honey comparator(1.5 tablespoons)
  Interventions: Dietary Supplement: Raw Honey; Dietary Supplement: Comparator

INTERVENTIONS:
Dietary Supplement: Raw Honey — Canada #2 white raw honey (1.5 tablespoons) supplied by SweetHeart Pollinators (Janeil Enterprises, Eatonia, SK) administered for 7 days
Dietary Supplement: Comparator — Honey comparator(1.5 tablespoons) administered for 7 days

SUMMARY:
Inadequate sleep quality and duration affects quality of life, and can cause adverse health outcomes, for many Canadians. Existing sleep therapies have limitations, such as inability to adhere to a cognitive behaviour modification or the risk of dependence on pharmaceutical therapies. Raw honey has a long history of anecdotal reports supporting its use to improve sleep quality. In an effort to develop an evidence base for honey as a sleep aid, we completed a preliminary proof-of-principle study to assess feasibility and potential effectiveness of honey to improve sleep quality. Results of our preliminary study demonstrate that honey is safe and effective for improving quality of sleep with no associated adverse effects, as compared to melatonin. The current study design builds off the experiences of the preliminary trial and will add more scientific rigor to the evidence base we have started to build.

DETAILED DESCRIPTION:
Inadequate sleep quality and duration may result in adverse health outcomes and poorer quality of life. Research thus far identify interventions such as behavior modification and pharmaceuticals to aid sleep. According to Stats Canada (2007-2013 Canadian Health Measures Survey), despite these available interventions, roughly half of men and women (43% and 55%, respectively) aged 18-64 have difficulty falling or staying asleep; these results are similar to those reported in 2005. The lack of improvement in sleep might reflect important limitations with the current interventions; individuals with sleep disorders may find adherence to such interventions difficult to maintain (e.g. behavior modification) or the therapies may pose a risk (e.g. dependence on pharmaceuticals). There is a clear need for alternative therapeutic interventions, particularly those that are simple and cost effective.

Observational and anecdotal evidence supports honey as an alternative to promote better sleep. During sleep, the brain typically utilizes liver glycogen stores to provide continuous and adequate energy; foods that promote liver glycogen storage before sleep may ensure availability of this energy source and therefore lead to better sleep.4 Raw honey is a rapidly digestible and metabolizable dense energy source, and thus may provide this sleep time energy reserve. Additionally, honey may promote melatonin formation due to its possible tryptophan content (a precursor to melatonin) that both helps to initiate sleep as well as promote release of hormones that facilitate whole body recovery during sleep.

Based on this information, we completed a preliminary open-label proof-of-principle study to assess the feasibility and potential effectiveness of honey in improving sleep quality. In a cross-over study of poor sleepers, honey improved some areas of sleep compared to melatonin. The results of this study are the driving factor for the randomized, double-blind, cross-over study in poor sleepers proposed here.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 - 55yrs
* Male or female
* Able to comply with study protocol and give informed consent
* Healthy (no diagnosis of medical or mental illness and not suffering from vascular disease, diabetes mellitus, hyperlipidemia, obesity [body mass index over 30], dermatological disease, gynecological disease, endocrine disease)
* Discontinuation of sleep aids 4 weeks in advance of the study
* Self-report of having difficulty sleeping for 1 week or more

Exclusion Criteria:

* Age: <18 and >55
* Type I and Type II diabetes, current infectious disease (e.g. cold or flu)
* Unstable medical condition
* History of psychiatric disorder (past or present)
* Pain syndrome affecting sleep
* Obese (BMI over 30)
* Pregnant or lactating women
* Lifestyle habits that would modify the wake-sleep rhythm (e.g. night work; shift work; young children that interrupt sleep)
* Substance and/or drug dependence (alcohol, nicotine, pain killers)
* Use of the following medications during the study period: oral or injectable corticosteroid, sedating antihistamines (e.g. cold, allergy, motion sickness), psychotropic medications or hypnotics, benzodiazepine, narcotics, any illicit drugs
* Use of stimulants (>4 cups [1 cup = 250 mL] of coffee/day)
* Participation in any other clinical trial with an investigational agent within one month prior to randomization

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Sleep quality as measured by Leeds Sleep Evaluation Questionnaire | 14 days
  Assessment of the quality of sleep as measured by a standardized tool, the Leeds Sleep Evaluation Questionnaire, which assesses subjective measures of sleep quality and amount, by the end of the 7 day intervention with the treatments (honey or comparator)

SECONDARY OUTCOMES:
Sleep quality as measured by daily sleep hygiene logs | 14 days
  Assessment of the quality of sleep as measured by a daily sleep hygiene log, which assesses subjective measures of sleep quality and amount by the end of the 7 day intervention with the treatments (honey or comparator)
Sleep quality as measured by daily morning sleep logs | 14 days
  Assessment of the quality of sleep as measured by a daily morning sleep log, which assesses subjective measures of sleep quality and amount by the end of the 7 day intervention with the treatments (honey or comparator)
Sleep quality as measured by actigraphy | 14 days
  Assessment of the quality of sleep as measured by actigraphy, which assesses objective measures of sleep quality and amount by the end of the 7 day intervention with the treatments (honey or comparator)

CONTACTS AND LOCATIONS:
Overall Officials: Jane Alcorn, PhD, Principal Investigator — University of Saskatchewan
Locations (1):
- University of Saskatchewan, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No